CLINICAL TRIAL: NCT04683952
Title: Efficacy of Exercise Training With Humified High Flow Nasal Cannula, in Patients With Chronic Obstructive Pulmonary Disease Already in Nocturnal Non-Invasive Ventilation
Brief Title: Rehabilitation With HHFNC in COPD in Nocturnal NIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDG_HFNC_COPD_01
Record Dates: First submitted 2020-05-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; HHFNC; Chronic Obstructive Pulmonary Disease; Humidified High Flow Nasal Cannula; Non Invasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation with HHFNC (Experimental): 15 Chronic Obstructive Pulmonary Disease patients in nocturnal Non Invasive Ventilation (NIV) who will perform rehabilitation, with / without Oxygen Therapy according to prescription, and with Humified High Flow Nasal Cannula (HHFNC).
  The Rehabilitation program consists in 20 session of 40 minutes, thrice a week for three times with a washout period of 3 months.
  Interventions: Device: Exercise training with Humified High Flow Nasal Cannula
- Control Group rehabilitation without HHFNC (Active Comparator): 15 Chronic Obstructive Pulmonary Disease patients in nocturnal Non Invasive Ventilation (NIV) who will perform rehabilitation, with / without Oxygen Therapy according to prescription, without Humified High Flow Nasal Cannula (HHFNC).
  The Rehabilitation program consists in 20 session of 40 minutes, thrice a week for three times with a washout period of 3 months.
  Interventions: Other: Exercise training - Control Group

INTERVENTIONS:
Device: Exercise training with Humified High Flow Nasal Cannula — The experimental group will be trained using HHFNC with the most adequate continuous flow, in a range between 25 and 30 L / min.
  Other Names: VEMO 150
  Arms: Rehabilitation with HHFNC
Other: Exercise training - Control Group — The control group will perform exercise training in spontaneous breathing.
  Arms: Control Group rehabilitation without HHFNC

SUMMARY:
Humidified High Flow Nasal Cannula (HHFNC), with optional supplemental oxygen delivery, has evolved in recent years with an increasing number of papers that show a better meet with respiratory demand, decrease oxygen dilution, increased Functional Residual Capacity (FRC), dead space washout, more tolerate than Non Invasive Ventilation (NIV) and provide heated and humidified gas. HHFNC is mainly used in intensive care settings or in acute respiratory diseases for the treatment of mild to moderate acute hypoxic respiratory failure and ventilator weaning. The aim of this study is to evaluate, in patients with Chronic Obstructive Pulmonary Disease (COPD) in nocturnal NIV, according to the European Respiratory Society (ERS) and American Thoracic Society (ATS) guidelines, whether HHFNC during rehabilitation has an additional effect in increasing the distance in 6 Minute Walking Distance (6MWD) compared to the control group with nocturnal NIV without HHFNC treatment. As secondary objectives, we expect a decrease in Emergency Department (ED) accesses, General Practitioner (GP) unplanned visits, hospitalizations and an improvement of the quality of life and patient satisfaction.

DETAILED DESCRIPTION:
RECRUITMENT PHASE: A qualified physiotherapist will check patient lists daily with the aim of identifying suitable candidates for the study.

The patients will be enrolled from January 2020 till june 2021 and they will be stratified individually and randomized by a dedicated software (https://www.randomizer.org/) into two groups:

* Experimental group - Chronic Obstructive Pulmonary Disease (COPD) patients in nocturnal Non Invasive Ventilation (NIV) underwent to respiratory rehabilitation with Humidified High Flow Nasal Cannula (HHFNC) with / without Oxygen Therapy (O2), according to medical prescription;
* Control group - patients in nocturnal NIV underwent to respiratory rehabilitation without HFNC with / without O2, according to medical prescription.

Before randomization, individual clinical inclusion and exclusion criteria will be taken into account in relation to the ability of each patient to tolerate the administration of the high flow ventilation program foreseen by the study.

RUN IN PHASE: After the assessment, each patient will perform a training session prior to the cycle ergometer, during which the subject will work on the workload and the established flow. The intensity of the workload will be 60-80% of the Wmax, calculated with the Hill's formula:

Wmax = ( 0.122 x 6MWD) + (72, 683 x Height) - 117.109

(where 6MWD is the distance walked on the 6-minute walk test, and the patient's height must be expressed in meters).

NIV and HHFNC will be administered through VEMO 150 (EOVE SA. 64000 Pau - France), a device with which it is possible setting up to 4 different ventilation programs. The High Flow can be delivered, as a continuous flow through the humidified nasal cannulas, up to 60 L / min with or without additional oxygen therapy according to medical prescription. The patients of the experimental group will be trained with the most adequate continuous flow, in a range between 20 and 60 L/min, according to the maximum flow supported by the patient.

FOLLOW UP PHASE: Outpatient rehabilitation will be performed in 3 cycles, each cycle in 40-minute sessions, 3 times a week. Each session starts with the cycle ergometer with a 5-minute warm-up to an intensity of 0 watts, continues with a 30-minute resistance training phase at a continuous target intensity (60-80% Wmax), then a warm-down of 5 minutes at an intensity of 0 watts.

The rehabilitation will be followed by a three-month washout period, for 3 cycles.

MEASUREMENTS: We have identified four periods to evaluate gas exchange, Forced expiratory volume in one second (FEV1) and respiratory muscle strength, dyspnea, exercise capacity, the presence of obstructive/central sleep apnea, prediction of mortality, activities of daily life, the impact of the disease and the quality of life.

These four periods are:

* T0: baseline;
* T1: at the end of the first rehabilitation cycle;
* T2: at the end of the second rehabilitation cycle;
* T3: at the end of the third rehabilitation cycle.

At the beginning of the study, demographics and clinical characteristics of eligible study participants will be collected.

Patients will be evaluated for:

* Blood gas analysis (BGA) in T0, T1, T2, T3;
* Spirometry: Forced Vital Capacity (FVC), FEV1 and FEV1/FEVC% in T0, T3;
* Questionnaire of the British Medical Research Council (MRC) modified, in T0, T1, T2, T3;
* Basic / Transition Dyspnea Index (BDI / TDI), in T0, T1, T2, T3;
* 6 Minute Walking Distance (6MWD) with / without oxygen therapy, according to the medical prescription during the effort, in T0, T1, T2, T3;
* COPD Assessment Test (CAT) in T0, T1, T2, T3;
* Night time Polygraph to detect apnea/hypopnea, in T0, T3 ;
* BODE INDEX (where BODE means body mass index, obstruction of air flow, dyspnoea and exercise capacity), in order to estimate the probability of survival, in T0, T1, T2, T3;
* Saint George Respiratory Questionnaire (SGRQ) to investigate the quality of life in T0 and T3;
* Evaluation of the perception of muscle fatigue and dyspnea (Borg RPE) and Visual Analogue Scale (VAS) each session.

During training, and the run-in phase, the physiotherapist will take note of FiO2 and of the dyspnea at the beginning and end of the session through VAS / BORG and again when the patient will be evaluated in 6MWD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) / Forced Vital Capacity (FVC) <0.7) ;
* Nocturnal Non Invasive Ventilation (NIV) prescription according to ATS/ERS guidelines with or without long-term oxygen therapy;
* Clinical stability (no exacerbation and no changing in respiratory drugs in the last 7 days);

Exclusion Criteria:

* Orthopedic or neurological pathologies that limit physical performance;
* Cognitive impairment (Mini-Mental State Examination <24);
* Advanced heart disease, pulmonary fibrosis, participation in other clinical studies in the six months preceding the start of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 6MWD | "Baseline ( pre-intervention)" and "Immediately after the intervention".
  The first outcome we expect to find is a change in the distance at 6-Minute Walking Distance (6MWD).

SECONDARY OUTCOMES:
Number of Exacerbations, GP visits and admission to ED and ICU | Through study completion, an average of 1 year.
  The second outcome is change of COPD exacerbation as admission to the Intensive Care Unit (ICU), to the admission to the ED with/without hospitalization, Generale Practitioner (GP) unplanned visits.

OTHER OUTCOMES:
Points at Saint George Respiratory Questionnaire (SGRQ) | "Baseline ( pre-intervention)" and "Immediately after the intervention".
  The third outcome concerns the quality of life for which we expect changes in the results at the Saint George Respiratory Questionnaire (SGRQ) in the experimental group. SGRQ: from 0 (no health impairment) to 100 (maximum health impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Banfi, MD, Principal Investigator — Fondazione Don C. Gnocchi - I.R.C.C.S. Santa Maria Nascente; Laila Di Pietro, RT, Study Chair — Fondazione Don C. Gnocchi - I.R.C.C.S. Santa Maria Nascente
Locations (1):
- IRCCS Santa Maria Nascente, Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwabbauer N, Berg B, Blumenstock G, Haap M, Hetzel J, Riessen R. Nasal high-flow oxygen therapy in patients with hypoxic respiratory failure: effect on functional and subjective respiratory parameters compared to conventional oxygen therapy and non-invasive ventilation (NIV). BMC Anesthesiol. 2014 Aug 7;14:66. doi: 10.1186/1471-2253-14-66. eCollection 2014. PMID 25110463
- [Background] Stephan F, Berard L, Rezaiguia-Delclaux S, Amaru P; BiPOP Study Group. High-Flow Nasal Cannula Therapy Versus Intermittent Noninvasive Ventilation in Obese Subjects After Cardiothoracic Surgery. Respir Care. 2017 Sep;62(9):1193-1202. doi: 10.4187/respcare.05473. Epub 2017 Aug 14. PMID 28807988
- [Background] Hill K, Jenkins SC, Cecins N, Philippe DL, Hillman DR, Eastwood PR. Estimating maximum work rate during incremental cycle ergometry testing from six-minute walk distance in patients with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2008 Sep;89(9):1782-7. doi: 10.1016/j.apmr.2008.01.020. PMID 18760164
- [Background] Ergan B, Oczkowski S, Rochwerg B, Carlucci A, Chatwin M, Clini E, Elliott M, Gonzalez-Bermejo J, Hart N, Lujan M, Nasilowski J, Nava S, Pepin JL, Pisani L, Storre JH, Wijkstra P, Tonia T, Boyd J, Scala R, Windisch W. European Respiratory Society guidelines on long-term home non-invasive ventilation for management of COPD. Eur Respir J. 2019 Sep 28;54(3):1901003. doi: 10.1183/13993003.01003-2019. Print 2019 Sep. PMID 31467119
- See also: The Global Initiative for Chronic Obstructive Lung Disease (GOLD) Global Strategy for the Diagnosis, Management and Prevention of Chronic Obstructive Pulmonary Disease — http://goldcopd.org/gold-reports/